CLINICAL TRIAL: NCT05662917
Title: What Are the Views of Palliative Care Patients Regarding the Use of Anticipatory Prescribing ?
Brief Title: Advance Care Planning in Palliative Care
Acronym: ANTICIPALL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0747; ID-RCB (Other: 2022-A02147-36)
Record Dates: First submitted 2022-12-12; First posted 2022-12-23 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Palliative Care
Keywords: Palliative care; Advance care planning; Anticipatory prescribing; End of life; Patient experiences
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Palliative care patients: * Palliative care patients
  * Suffering from a serious and progressive illness (whatever it is)
  * Hospitalized in a palliative care unit or followed at home by the hospital's mobile palliative care team
  Interventions: Behavioral: Individual semi-structured interviews

INTERVENTIONS:
Behavioral: Individual semi-structured interviews — After information and written consent, the investigator will interview the participants through a semi-structured individual interview (conducted by an interview guide). The interview is expected to last 45 minutes (variable depending on the subject). It will be recorded by dictaphone, respecting the anonymity of the participant throughout the interview. The subject's participation will end after the interview.

SUMMARY:
The question of the end of life is a major public health issue. In the field of palliative care, the notion of anticipation is central for people with a serious and progressive illness. Indeed, an important consideration for general practitioners is the need to anticipate the disease's evolution and the uncomfortable symptoms (physical or psychological) the patient is likely to experience. This approach aims to relieve the patient without delay and thus improve comfort to ensure an acceptable quality of life for patients and their families. Even if the usefulness of anticipatory prescribing seems obvious, their use is not generalized to all palliative care patients. Caregivers are confronted with obstacles to the implementation of these prescriptions, particularly with regard to the relationship with the patient. It can then be assumed that patients' experiences and perceptions may influence symptom management and the use of anticipatory prescriptions. It seems essential to explore this subject. For this purpose, the investigator will carry out a qualitative study based on individual semi-structured interviews with palliative care patients.

ELIGIBILITY:
Inclusion Criteria:

* Persons of all genders
* Persons 18 years of age and older
* In a palliative care situation of any serious illness
* Persons hospitalized in palliative care unit at the Givors hospital or followed at home by the Mobile Palliative Care Team
* Patients who have received full information about the study and signed a written consent.

Exclusion Criteria:

* Persons under legal protection
* Persons unable to express their consent, making it impossible to conduct interviews: dysarthria, cognitive disorders, mental confusion, altered state of consciousness
* Pregnant or breastfeeding persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population concerns patients in palliative situation, either hospitalized in palliative care unit or followed at home by the Mobile Palliative Care Team. The number of subjects required is estimated at a minimum of 15 participants (depend on data saturation)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-12-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is patient views on the use of anticipatory prescribing. | The outcome will be collected at Day 1-End of study visit
  The interview consists in exploring the participants' experiences (feelings, representations), expectations and difficulties concerning the use of anticipatory prescribing. Interviews will be audio recorded. The verbatim will be transcribed for qualitative analysis by inductive thematic type, in order to bring out the main ideas and hypotheses.

CONTACTS AND LOCATIONS:
Overall Officials: Manon JULLIAN, Principal Investigator — Multidisciplinary medicine and palliative care department
Locations (1):
- Givors Hospital Center - Multidisciplinary medicine and palliative care department, Givors, France